CLINICAL TRIAL: NCT05963932
Title: A Phase 1, Open-label, Randomized, Parallel-group, Single Dose Study to Assess the Relative Bioavailability of a New BMS-986419 Immediate-release Tablet Formulation Compared to a Reference Enteric Capsule (Delayed-release) Formulation, and to Assess the Effect of Food on the Pharmacokinetics of Immediate-release Tablet Formulation in Healthy Adult Participants
Brief Title: A Study to Assess the Bioavailability and Effect of Food of BMS-986419 Immediate-release Tablet Formulation in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CN007-1001
Record Dates: First submitted 2023-07-20; First posted 2023-07-27 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Healthy Volunteers
Keywords: BMS-986419; Healthy male of non-child bearing potential; Healthy women of non-child bearing potential

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment A: BMS-986419 DR Capsule - Fasted (Experimental)
  Interventions: Drug: BMS-986419 DR Capsule
- Treatment B: BMS-986419 IR Tablet - Fasted (Experimental)
  Interventions: Drug: BMS-986419 IR Tablet
- Treatment C: BMS-986419 IR Tablet - Fed (Experimental)
  Interventions: Drug: BMS-986419 IR Tablet
- Treatment D: BMS-986419 Crushed IR Tablet - Fed (Experimental)
  Interventions: Drug: BMS-986419 IR Tablet

INTERVENTIONS:
Drug: BMS-986419 DR Capsule — Specified dose on specified days
  Arms: Treatment A: BMS-986419 DR Capsule - Fasted
Drug: BMS-986419 IR Tablet — Specified dose on specified days
  Arms: Treatment B: BMS-986419 IR Tablet - Fasted; Treatment C: BMS-986419 IR Tablet - Fed; Treatment D: BMS-986419 Crushed IR Tablet - Fed

SUMMARY:
The purpose of this study is to assess the impact of the BMS-986419 new immediate release (IR) tablet formulation compared to the current enteric (DR) capsule formulation, and to assess the effect of food on the drug levels of the IR tablet formulation in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female participants without clinically significant deviation from normal, as determined by the investigator, in medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory evaluations.
* Body mass index (BMI) of 18.0 to 32.0 kilograms per meter squared (kg/m^2), inclusive, and body weight ≥ 50 kg.
* A female participant is eligible to participate if she is a woman not of childbearing potential (WNOCBP)

Exclusion Criteria:

* Any significant acute or chronic medical illness (eg, history of intracranial or intraspinal hemorrhage, CNS lesions, recent bacterial or fungal meningitis, etcetera) as determined by the investigator.
* Current or recent (within 3 months of study intervention administration) gastrointestinal disease that could affect the absorption, distribution, metabolism, and excretion of study intervention (for example, bariatric procedure).
* History of Gilbert's syndrome.
* Women who are of childbearing potential and women who are breastfeeding.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-08-08 (Actual); Primary Completion 2023-10-17 (Actual); Study Completion 2023-10-17 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to 15 days
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUC [0-T]) | Up to 15 days
Area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUC[INF]) | Up to 15 days

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to 29 days
Number of participants with vital sign abnormalities | Up to 29 days
Number of participants with electrocardiogram (ECG) abnormalities | Up to 29 days
Number of participants with clinical laboratory abnormalities | Up to 29 days
Number of participants with physical examination abnormalities | Up to 29 days
Time to attain maximum observed plasma concentration (Tmax) | Up to 15 days
Terminal half-life (T-Half) | Up to 15 days
Area under the plasma concentration-time curve from time zero to 24 hours (AUC(0-24)) | Up to 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Anaheim Clinical Trials, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: No
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-andpartners/ clinical-trials-andresearch/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm